CLINICAL TRIAL: NCT04950933
Title: A Multi-center, Randomized, Double-blind, Positives Parallel Controlled, Phase Ⅱ Clinical Trial to Evaluate the Efficacy and Safety of Huollingshengji Granules in the Treatment of Amyotrophic Lateral Sclerosis (Spleen qi Deficiency, Kidney Yang Deficiency Syndrome)
Brief Title: The Treatment of Amyotrophic Lateral Sclerosis With Huollingshengji Granules
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2020076
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Drug: Huolingshengji Granules
- Control group (Placebo Comparator)
  Interventions: Drug: Riluzole tablet

INTERVENTIONS:
Drug: Huolingshengji Granules — 1 bag of Huolingshengji Granules each time + 1 tablet of Riluzole tablet simulation agent each time, twice a day, orally;
  Arms: Test group
Drug: Riluzole tablet — Huolingshengji granules simulation agent 1 bag each time + Riluzole tablet 1 tablet each time, 2 times a day, orally.
  Arms: Control group

SUMMARY:
This study intends to evaluate the efficacy and safety of Dong Lingsheng Ji Granule in the treatment of amyotrophic lateral sclerosis (spleen deficiency, kidney-yang deficiency syndrome) in comparison with riluzole, so as to provide data support for marketing application or subsequent clinical research design.

DETAILED DESCRIPTION:
This study proposed the multicenter, randomized, double-blind, double simulation, positive drug parallel contrast the bad effect of experimental design, into the treatment group 72 cases, control group of 72 cases with the azole comparison, evaluation Dong Ling raw grain treatment on muscle atrophy amyotrophic lateral sclerosis (lack of temper, kidney Yang deficiency syndrome) efficacy and safety, for applications or follow-up clinical study design to provide data support.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Western diagnostic criteria for amyotrophic lateral sclerosis (ALS) (clinically confirmed ALS, clinically likely ALS or clinically likely ALS- laboratory support);
2. The score of the modified amyotrophic lateral sclerosis function scale (ALSFRS-R) was ≥2 points for each item (among which dyspnea, sitting breathing and respiratory insufficiency were all 4 points);
3. The percentage of forced vital capacity in the predicted value (FVC%) ≥70%;
4. the duration of the disease is 3 years or less (from the first onset of any symptoms of ALS);
5. TCM syndrome differentiation for deficiency of temper, kidney Yang deficiency syndrome;
6. Age 45-70 (including 45 and 70), gender unlimited;
7. Voluntarily participate in the clinical trial, give informed consent and sign informed consent.

Exclusion Criteria:(1) Patients diagnosed with familial ALS; (2) Those who have undergone gastrostomy; (3) patients with other neurological diseases similar to ALS, such as cervical spondylotic myelopathy, lumbar spondylopathy, dementia, etc., which may affect the evaluation of drug effectiveness; (4) electromyogram detection found motor nerve conduction block, sensory nerve conduction abnormality, imaging examination (CT or MRI) found that can explain the clinical manifestations of substantial lesions; (5) Patients who had been treated with riluzole or edaravone within 3 months before enrollment; (6) patients with a history of spinal surgery after the onset of ALS; (7) aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times the upper limit of the normal reference value, or blood muscle (SCR) >; Upper limit of normal reference value; (8) Patients with other serious primary diseases of the nervous system, heart, lung, hematopoietic system or endocrine system and psychosis; (9) Suspected or have a history of alcohol and drug abuse; (10) Pregnant women or lactating women, subjects of reproductive age (including male subjects with heterosexual behavior and their female partners with fertility potential) have pregnancy plans or are unwilling to take effective contraceptive measures within 3 months from the beginning of screening to the end of drug withdrawal; (11) People who are known or suspected to have a history of allergy to the test drug and its excipients; (12) Screening participants who had participated in other clinical trials within the previous 3 months; (13) Those considered by the researcher to be unsuitable to participate in this clinical trial.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R scores | 48 weeks
  Changes in ALSFRS-R scores from baseline after 48 weeks of treatment, The ALSFRS-R scale (ALS Functional Rating Scale) includes 12 items including medulla oblongata function, limb function and respiratory function, with a total score of 48. The lower the score, the more serious the neurological function damage.

SECONDARY OUTCOMES:
FVC% | 48 weeks
  Change in FVC% from baseline after 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No